CLINICAL TRIAL: NCT00486551
Title: Anger Control Training for Youth With Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Tourette Association of America (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0102012121; 1R03MH067845 (NIH)
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Tourette Syndrome; Chronic Tic Disorder; Oppositional Defiant Disorder; ADHD
Keywords: Anger control training; Cognitive behavioral therapy; Behavior therapy; Tourette Syndrome; Randomized trial; Anger; Aggression
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Oppositional Defiant Disorder; Attention Deficit Disorder with Hyperactivity; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Anger control training

SUMMARY:
This is a clinical study of a cognitive-behavioral therapy known as anger control training in adolescents with Tourette Syndrome and explosive, disruptive behavior. ACT is compared to treatment as usual (TAU) in a randomized clinical trial.

DETAILED DESCRIPTION:
This is a randomized controlled study of a cognitive-behavioral, anger control training (ACT) in adolescents with Tourette Syndrome (TS) complicated by disruptive behavior. Disruptive behaviors in TS may take numerous forms including noncompliance, anger outbursts, and physical aggression. Anger outbursts in TS have been described as rage attacks or rage storms due to their high intensity and unpredictability in response to minimal provocation. Whether these behaviors are part of TS, related to comorbid conditions, or due to the burden of chronic illness is not clear. Nevertheless, these disruptive behaviors can result in significant functional impairment and often require clinical attention. The purpose of the ACT intervention is to improve the explosive and noncompliant behavior in adolescents with TS by enhancing affect regulation and social problem-solving skills. The treatment is based on anger control training which has been empirically supported for reducing aggressive behaviors and improving social functioning in aggressive youths. The primary outcome measures include the parent-rated Oppositional Defiant Scale and the Clinicians Global Improvement Score assessed by a clinician blind to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Boys and girls, 11 to 16 years of age.
2. Diagnosis of Tourette syndrome (TS) or chronic tic disorder (CTD).
3. Significant level of disruptive behavior

Exclusion Criteria:

1. Current diagnosis of Severe Major Depression, Bipolar Disorder, Pervasive Developmental Disorder, or Psychotic Disorder.
2. Significant medical condition such as heart disease, hypertension, liver or renal failure, pulmonary disease, seizure disorder that may require more pressing treatment.
3. Initiation or discontinuation of a psychotropic medication treatment within six weeks of enrollment in the study

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2001-08; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
CGI-I assigned by clinician unaware of treatment assignment | three months
Parent rated disruptive behavior | three months

CONTACTS AND LOCATIONS:
Overall Officials: Denis G Sukhodolsky, Ph.D., Principal Investigator — Yale University; Lawrence D Scahill, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Sukhodolsky DG, Scahill L, Zhang H, Peterson BS, King RA, Lombroso PJ, Katsovich L, Findley D, Leckman JF. Disruptive behavior in children with Tourette's syndrome: association with ADHD comorbidity, tic severity, and functional impairment. J Am Acad Child Adolesc Psychiatry. 2003 Jan;42(1):98-105. doi: 10.1097/00004583-200301000-00016. PMID 12500082
- [Background] Sukhodolsky DG, do Rosario-Campos MC, Scahill L, Katsovich L, Pauls DL, Peterson BS, King RA, Lombroso PJ, Findley DB, Leckman JF. Adaptive, emotional, and family functioning of children with obsessive-compulsive disorder and comorbid attention deficit hyperactivity disorder. Am J Psychiatry. 2005 Jun;162(6):1125-32. doi: 10.1176/appi.ajp.162.6.1125. PMID 15930061
- [Background] Scahill L, Erenberg G, Berlin CM Jr, Budman C, Coffey BJ, Jankovic J, Kiessling L, King RA, Kurlan R, Lang A, Mink J, Murphy T, Zinner S, Walkup J; Tourette Syndrome Association Medical Advisory Board: Practice Committee. Contemporary assessment and pharmacotherapy of Tourette syndrome. NeuroRx. 2006 Apr;3(2):192-206. doi: 10.1016/j.nurx.2006.01.009. PMID 16554257
- [Result] Sukhodolsky DG, Vitulano LA, Carroll DH, McGuire J, Leckman JF, Scahill L. Randomized trial of anger control training for adolescents with Tourette's syndrome and disruptive behavior. J Am Acad Child Adolesc Psychiatry. 2009 Apr;48(4):413-421. doi: 10.1097/CHI.0b013e3181985050. PMID 19242384
- See also: Related Info — http://childstudycenter.yale.edu/